CLINICAL TRIAL: NCT06671730
Title: Digitally Mediated Occupational Therapy Program to Increase Physical Activity in Urban and Rural Breast Cancer Survivors Who Have Undergone Breast-conserving Surgery or Mastectomy
Brief Title: Self-Determination Theory-informed Occupational Therapy Program to Increase Physical Activity Among Survivors of Breast Cancer
Acronym: SDOTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16601; IRG-23-1143225-04-IRG (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Survivor
Keywords: Aerobic Physical Activity; Muscle Strengthening Exercise; Patient Reported Outcomes; Feasibility; Acceptability; Wearable Devices; Telehealth

STUDY DESIGN:
Intervention Model Description: We will investigate the acceptability and feasibility of a novel 8-week occupational therapy (OT) program among 38 rural and urban breast cancer (BC) survivors that features: 1) 8 weekly telehealth OT sessions, and 2) self-regulatory strategies known to support aerobic physical activity (PA) and muscle strengthening exercise (MSE) adoption and maintenance, emphasizing components of the Self-Determination Theory (SDT), and the provision of a wearable device (e.g., a fitness tracker) programmed to supplement individually tailored goals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 8-Week Telehealth-delivered Occupational Therapy Program (Experimental): The telehealth-based OT program will be grounded in SDT. The program will be designed to help BC survivors transition from recovery after surgery to achieving levels of aerobic PA and MSE that are recommended according to each participants' specific treatment course and desired outcomes. Participants will engage in eight once-weekly OT sessions with a licensed occupational therapist via Zoom-lasting for up to about an hour. Each session will teach psychoeducational and skill-building techniques that support decreasing functional limitations associated with BC and BC treatment as well as improving behavioral skill sets necessary for maintenance of aerobic PA and MSE. Participants will receive study-provided exercise equipment and a fitness tracker (Fitbit Charge 6) for use engaging in greater amounts of aerobic PA and MSE (keeping these materials post-study).
  Interventions: Behavioral: 8-Week Telehealth-based Occupational Therapy Program

INTERVENTIONS:
Behavioral: 8-Week Telehealth-based Occupational Therapy Program — The telehealth-based OT program will be grounded in SDT. The program will be designed to help BC survivors transition from recovery after surgery to achieving levels of aerobic PA and MSE that are recommended according to each participants' specific treatment course and desired outcomes. Participants will engage in eight once-weekly OT sessions with a licensed occupational therapist via Zoom-lasting for up to about an hour. Each session will teach psychoeducational and skill-building techniques that support decreasing functional limitations associated with BC and BC treatment as well as improving behavioral skill sets necessary for maintenance of aerobic PA and MSE. Participants will receive study-provided exercise equipment and a fitness tracker (Fitbit Charge 6) for use engaging in greater amounts of aerobic PA and MSE (keeping these materials post-study)

SUMMARY:
We will evaluate a novel 8-week telehealth-delivered occupational therapy (OT) program among breast cancer survivors that seeks to promote engagement in aerobic physical activity (PA) and muscle strengthening exercise (MSE). The telehealth-based delivery of this OT program circumvents some barriers to OT access and participation (e.g., time burden; distance to OT clinic) among breast cancer survivors- particularly important for Oklahoma given that 33% of residents live in rural areas. Additionally, the focus of this program is to promote the preferred aerobic PA and MSE choices of each individual survivor to increase the likelihood of long-term PA engagement. In turn, participants will be more likely to experience the longer-term benefits associated with PA such as improved physical functioning, reduced anxiety, depressive, and pain symptoms, better sleep, and better cardiorespiratory fitness.

DETAILED DESCRIPTION:
Breast cancer (BC) survivors, defined as those ever diagnosed with BC through the end of life, totaled approximately 4 million people in the U.S. in 2022. While the 5-year survival rate across all races for BC is 90%, functional limitations associated with BC treatment often have considerable impacts on BC survivors' physical and mental health-related quality of life (HRQoL). Approximately 90% of women diagnosed with non-metastatic BC undergo breast-conserving surgery or mastectomy. These surgical interventions commonly lead to upper extremity impairment, decreased strength, and limited mobility, contributing to long-term declines in objectively measured physical function, one key determinant of HRQoL. Moreover, BC survivors' functional limitations can limit participation in health promoting behaviors (e.g., aerobic physical activity [PA]; muscle strengthening exercise [MSE])-limitations that have been shown to place this population at increased morbidity and premature mortality risk. It is therefore critical to develop accessible programs that allow BC survivors who have undergone breast-conserving surgery or mastectomy to reduce functional limitations and more readily engage in health promoting behaviors contributing to improved HQRoL.

Physical activity is safe and beneficial for most cancer survivors, and can improve HRQoL via increased self-efficacy and physical, emotional, social, and functional well-being. More specifically, aerobic PA has been shown to have a positive impact on multiple aspects of BC survivors' health, including cardiorespiratory fitness and fatigue levels. Recently, MSE has been established as a critical health-promoting behavior for reducing the functional limitations associated with BC treatment. MSE also contributes to improved cardiorespiratory fitness and overall metabolic health. However, less than 20% of BC survivors meet recommended aerobic PA and MSE guidelines. Qualitative research highlights that BC survivors who have undergone breast-conserving surgery or mastectomy are uncertain about integrating aerobic PA and MSE into their lives after transitioning out of formal care settings. Support is needed to help this population with lingering functional limitations transition into sustained, self-directed PA and MSE in community- and home-based settings.

Occupational therapy (OT) is uniquely capable of addressing the barriers to sustained PA faced by BC survivors who have undergone breast-conserving surgery or mastectomy. The goal of OT for cancer survivors is to return to activities of daily living following cancer treatment. As such, OT is a critical post-treatment component for BC survivors. Occupational therapists are trained in behavior change techniques, remediation of functional impairments, and modification of activities and environments. This training uniquely positions occupational therapists to provide the specialized aerobic PA and MSE programming that can support BC survivors' health behavior initiation and maintenance. Further, this skillset may be particularly conducive to promoting long-term adherence to aerobic PA and MSE, as OT emphasizes the primacy of building clients' capacity to engage in behaviors that are congruent with personally held values and preferences. Emerging evidence suggests that orienting health promotion efforts in this way supports sustained lifestyle behavior change.

OT-based PA programming for BC survivors can be grounded in Self-Determination Theory (SDT) to support sustained, self-directed PA. SDT posits that people are oriented toward growth and development, and that the satisfaction of people's core psychological needs (i.e., autonomy, competence, and relatedness) facilitates the formation of autonomous motivations for health-related behaviors (i.e., enjoyment, interest, identity, and values). It theorizes that changes in more autonomous motivations will yield longer-lasting behavioral changes than changes in less autonomous motivations. Autonomous motivations for PA are well established determinants of long-term physical activity maintenance in multiple populations, including BC survivors. Autonomous motivations for PA can be modified by targeting core psychological needs (i.e., increasing perceptions of autonomy, competence, and relatedness). Importantly, SDT has been proposed as an ideal theoretical framework for guiding OT. OT is centered on building client's capacity to engage in personally defined goals and occupations (targeting perceptions of autonomy). Occupational therapists scaffold learning and apply therapeutic techniques centered on helping clients experience incremental successes toward achieving their goals (competence); they also prioritize establishing an autonomy-supportive, therapeutic alliance with their clients (relatedness). It is through these mechanisms of action that we expect our program to yield sustained increases in aerobic PA/MSE for BC survivors.

Digitally mediated occupational therapy (OT) is uniquely suited to helping BC survivors transition to sustained community- and home-based physical activity after undergoing breast surgery dramatically increasing the accessibility of expert-provided PA/MSE programing. OT programs conducted in formal settings are often associated with low adherence and face marked barriers to implementation, including lack of access to care and transportation-related barriers. These barriers are most pronounced in rural BC survivors-particularly relevant to the target population of the current proposal; in 2020, 33% of Oklahomans lived in areas designated as 'rural' by the U.S. Department of Agriculture (USDA) Economic Research Service (ERS). The use of digital technologies, such as telehealth, can help rural and urban BC survivors circumvent these challenges to receiving OT programming. Emerging evidence suggests that technology-mediated OT is feasible for urban and rural BC survivors. Yet, more research is needed to understand if a telehealth-delivered OT program based on the tenets of SDT and focused on promoting post-surgery aerobic PA and MSE will be acceptable and feasible to urban and rural BC survivors. We propose to investigate the acceptability, feasibility, and safety of a novel 8-week OT program among urban and rural BC survivors (N = 30) that combines 1) 8 telehealth-delivered sessions with an occupational therapist and 2) self-regulatory strategies known to support PA adoption and maintenance.1 Study observations will contribute valuable insights regarding how to scale telehealth-delivered OT programs to improve PA adherence and PROs among urban and rural BC survivors-ultimately helping improve HRQoL.

We will investigate the acceptability and feasibility of a novel 8-week OT program among 30 rural and urban BC survivors that features: 1) 8 weekly telehealth OT sessions, and 2) self-regulatory strategies known to support aerobic PA and MSE adoption and maintenance, emphasizing components of the SDT, and the provision of a wearable device (e.g., a fitness tracker) programmed to supplement individually tailored goals. We have the following Specific Aims, Hypotheses, and Milestones:

Aim 1: Assess participants' perceptions of the acceptability, usability, and usefulness of the SDT-grounded, OT-based PA/MSE program (hereafter 'program'). Hypothesis 1: Participants will report the program's components to be acceptable, useable, and useful. Milestone 1a: Thematic analyses of qualitative data will suggest the program was enjoyable and improved physical and mental well-being. Milestone 1b: Quantitative assessments of the program via the System Usability Scale will average scores >68-indicative of 'above-average' program usability and usefulness.

Aim 2: Evaluate program feasibility and safety. Hypothesis 2: The program will be feasible and safe as demonstrated by satisfactory participant retention and adherence to program components and no unexpected increases in adverse outcomes. Milestone 2a: At least 80% of participants who complete baseline measures will subsequently complete post-program measures Milestone 2b: Participants will average ≥80% attendance at OT sessions. Milestone 2c: Frequency of BC-related lymphedema, musculoskeletal injuries, and any adverse events will be below normative values-indicative of a safe program.

Exploratory Aims: Evaluate pre- to post-program changes in 1: SDT-related constructs as key mechanisms of action; 2: aerobic PA and MSE; and 3: patient-reported outcomes (PROs) and goal attainment. Exploratory Hypotheses: Pre- to post-program changes in SDT-related components, aerobic PA and MSE behaviors, and PROs/goal attainment will be favorable. Milestone 3a: Measures of perceived autonomy, competence, and relatedness-key SDT components in the context of PA/MSE-will improve from pre- to post-program. Milestone 3b: Participants will demonstrate aerobic PA increase of ≥10 minutes/day and will engage in at least two MSE bout per week by post-program. Milestone 3c: An average pre- to post-program change of 2-6 T-score points, dependent on the PRO being assessed, as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS), with most participants achieving their pre-program goals by post-program.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old.
2. Ability to speak/read English.
3. Ability to provide informed consent.
4. Having ever received a histologically confirmed diagnosis of invasive breast carcinoma.
5. Having undergone breast conserving surgery or mastectomy for BC in the last 12 months.
6. Owning a smartphone and/or computer with internet access.
7. Willing to participate in once-weekly telehealth-delivered OT sessions for eight weeks.

Exclusion Criteria:

1. Currently undergoing chemotherapy or radiation as primary cancer treatment.
2. Planning or preparing for surgery as primary treatment or as a reconstruction procedure in the next 3 months.
3. Presence of distant metastasis.
4. Reporting a Physical Activity Readiness Questionnaire (2017 PAR-Q+) score that indicates PA may potentially be unsafe, unless the participant produces a signed doctor's note. We will define 2017 PAR-Q+ scores as indicating that PA may potentially be unsafe as responding "Yes" to any of the follow-up questions except [1] if the individual indicates that they have high blood pressure but subsequent responses indicate that both they do not have problems keeping it under control and that their resting blood pressure is less than 160/90 mmHg, and [2] if the individual indicates that they have a metabolic condition but subsequent responses indicate that they do not have problems controlling their blood sugar levels, do not any experience signs or symptoms of hypoglycemia, and do not have any signs of symptoms of listed diabetes complications).
5. Already engaging in ≥ 75 min/week of vigorous-intensity PA, ≥ 150 min/week of moderate-intensity PA, or an equivalent combination of both over the last 3 months.
6. Being a prisoner, pregnant, or planning to become pregnant.
7. Currently participating in another PA- or OT-based study, or seeking physical therapy or occupational therapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-17 (Estimated)

PRIMARY OUTCOMES:
Program Acceptability | End of Study Week 8
  Semi-structured Interviews and face valid questionnaires will be used to determine whether BC survivors found the intervention acceptable. The semi-structured interviews will be evaluated via thematic analysis, and the questionnaires will be scored on a 7-point Likert scale (1: 'Not at all'; 7: 'Very'), with higher scores being better.
Program Usability | End of Study Week 8
  Semi-structured interviews and face valid questionnaires will be used to determine whether BC survivors found the intervention useful as well as how it could be improved in the future. The semi-structured interviews will be evaluated via thematic analysis, and the questionnaires will be scored on a 7-point Likert scale (1: 'Not at all'; 7: 'Very'), with higher scores being better.
Program Usefulness | End of Study Week 8
  Semi-structured Interviews and face valid questionnaires will be used to determine whether BC survivors found the intervention useful at helping them increase their ability to engage in PAs that they value most. The semi-structured interviews will be evaluated via thematic analysis, and the questionnaires will be scored on a 7-point Likert scale (1: 'Not at all'; 7: 'Very'), with higher scores being better.

SECONDARY OUTCOMES:
Feasibility: Program Recruitment | From Baseline through Study Week 8
  Recruitment rates will be reported as the proportion of BC survivors enrolled in the study divided by the number of BC survivors who complete the screening survey. Enrollment will be considered feasible if ≥70% of eligible and approached BC survivors consent and enroll.
Feasibility: Program Retention | From Baseline through Study Week 8
  Study retention will be the number of BC survivors completing the program divided by the number that started. Retention will be considered feasible if ≥80% BC survivors who complete the baseline measures also complete measures post-program.
Feasibility: Program Adherence | From Baseline through Study Week 8
  The number of weekly telehealth-delivered OT sessions (out of eight total sessions) that each participant attends will be used as the program adherence metric. Adherence will be considered feasible if participants average ≥80% attendance OT sessions.
Program Safety: Incidence of Lymphedema Events, Musculoskeletal Injuries, and Adverse Events | From Baseline through Study Week 8
  Assessments of program safety will be assessed by tracking any BC-related lymphedema events, musculoskeletal injuries, and adverse events. The occupational therapist will track this information each week during each participant's telehealth-delivered OT session. The program will be considered safe if these events occur at or below published normative values.

OTHER OUTCOMES:
Psychological Needs Satisfaction | From Baseline through Study Week 8
  We will assess participants' pre- to post-program changes in SDT constructs through examinations of basic psychological needs satisfaction in exercise. We will operationalize these constructs using the Basic Psychological Needs in Exercise Scale. This 11-item Likert-type scale that features three subscales that measure perceptions of autonomy, competence, and relatedness (1: "I don't agree at all"; 5: "I completely agree").
Theory Intervention Fidelity Test | End of Study Week 8
  This measure will allow us to assess participants' perceptions of having experienced the SDT's underlying mechanisms of behavior change (autonomy, competence, and relatedness) as well as meaning associated with the intervention's aim (i.e., to increase engagement in personally meaningful physical activities). Responses are on a 7-point Likert-type scale (1: "Strongly disagree"; 7: "Strongly agree"), with higher scores better.
Supportive Accountability Inventory | End of Study Week 8
  The Supportive Accountability Inventory will allow us to assess the degree of supportive accountability participants felt the study occupational therapist provided during the course of the program. Participants will respond on a 7-point Likert scale (1 = 'Strongly disagree; 7 = 'Strongly agree').
Physical Activity | During the Baseline Week and Study Week 9
  Measurements of pre- to post-program changes in aerobic PA will be completed using ActiGraph GT3X accelerometers. Durations of moderate-vigorous physical activity [MVPA], light physical activity [LPA], and sedentary behavior (SB) reported will aggregated and reported as our single overall physical activity metric.
MSE Bouts | From Baseline through Study Week 8
  Pre- to post-program changes in weekly MSE bouts will be tracked as the occupational therapist discusses PA goals with each participant during their once-weekly OT session. The occupational therapist's notes will be used to determine the percentage of program weeks that BC survivors meet the recommended two bouts of MSE per week.
Health-related Quality of Life | Baseline and End of Study Week 8
  We will evaluate pre- to post-program changes in HRQoL using patient-reported outcomes. We will assess the following eight components of physical and psychological health at baseline and post-program using the Patient-Reported Outcomes Measurement Information System (PROMIS): physical functioning, fatigue, anxiety, depression, pain interference, pain intensity, sleep impairment, and sleep disturbance. Measurements on the PROMIS are on a 5-point Likert-type scale, with 5 reflecting worse outcomes on all components aside from physical function wherein a higher score reflects better physical function. These PROMIS measures have been observed as reliable tools for the assessment of these outcomes.
Goal Attainment | From Baseline through Study Week 8
  We will measure Goal attainment via goal attainment scaling (GAS). Measurement/Analysis: GAS allows for reporting the extent to which a participant meets weekly goals using a 5-point scale (-2 [minimum]: performance was much worse than expected; +2 [maximum]: performance was much better than expected). Measurement of pre-post changes obtained through transforming into a single aggregate score using established protocols.
Sociodemographics and Health History | Baseline
  We will collect social and demographic variables at baseline to ensure we can best describe our sample and explain observation nuances (e.g., age, sex, race/ethnicity, education, height and weight, marital status, annual household income, date of BC diagnosis and stage at diagnosis, type of BC treatment(s) received, comorbidities [e.g., type II diabetes], readiness to change, and overall health status).

CONTACTS AND LOCATIONS:
Overall Officials: Tara C Klinedinst, PhD, Principal Investigator — University of Oklahoma Health Sciences; Michael C Robertson, PhD, MPH, Principal Investigator — University of Oklahoma Health Sciences; Zachary C Pope, PhD, Principal Investigator — University of Oklahoma Health Sciences
Locations (1):
- University of Oklahoma Health Sciences, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Klinedinst TC, Pope ZC, Robertson MC, Stanley N, Wint A, Henson C, Kendzor DE. Digitally Mediated Occupational Therapy to Increase Physical Activity in Urban and Rural Breast Cancer Survivors: Protocol for a Single-Arm Feasibility Trial. JMIR Res Protoc. 2025 Sep 26;14:e73554. doi: 10.2196/73554. PMID 41004800